CLINICAL TRIAL: NCT01953861
Title: An Open-label, Single Dose, Randomized, Three-way Cross-over Study to Evaluate the Effect of Food on the Pharmacokinetics of Solifenacin and Tamsulosin Administered as Combination Tablet EC905 in Young, Healthy Male Subjects
Brief Title: A Study to Evaluate Whether Food Has an Effect on the Uptake of Solifenacin and Tamsulosin When Administered in a Combination Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 905-CL-054; 2009-013419-36 (EudraCT Number)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: EC905; Pharmacokinetics; Healthy Subjects
Keywords: Phase I; Combination tablet EC905; Omnic OCAS®; Vesicare®; Food effect; Vesomni; VesiFlow; Urizia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1: fasted (Experimental): EC905 + fasted
  Interventions: Drug: EC905
- 2: low-fat breakfast (Experimental): EC905 + low-fat breakfast
  Interventions: Drug: EC905
- 3: high-fat breakfast (Experimental): EC905 + high-fat breakfast
  Interventions: Drug: EC905

INTERVENTIONS:
Drug: EC905 — Oral
  Other Names: Vesomni; VesiFlow; Urizia

SUMMARY:
To evaluate the effect of food (low and high fat breakfast vs. fasting) on the pharmacokinetics (what the body does to the drug) of a single dose of solifenacin and tamsulosin administered as combination tablet EC905. Also to evaluate the safety and tolerability of single doses of EC905 in young, healthy male subjects, when administered under fed (low and high fat) or fasting conditions.

DETAILED DESCRIPTION:
Subjects are admitted to the clinic on Day -1 and receive a single dose of the combination tablet EC905 on the first day of 3 periods, under three conditions (high fat breakfast, low fat breakfast, and fasting) in order to evaluate the effect of food.

Blood sampling for pharmacokinetic (PK) assessment is performed on the dosing day and for 11 days after dosing in each period. This 11-day on-site period is repeated three times so that all subjects are dosed under all conditions. Each period is separated by 7 days off site.

Subjects return for an End of Study Visit (ESV) at least 7 days after the last 11 day on-site period, or after withdrawal.

On Day 1 of each of 3 periods, subjects are given a single dose of EC905 under three conditions (high fat breakfast, low fat breakfast and fasting) in order to evaluate the effect of food on the PK of solifenacin and tamsulosin HCl. The aim is to show the absence of a food effect after a low fat breakfast vs. fasting conditions, and to evaluate the food effect after a high fat breakfast vs. fasting conditions.

Subjects are randomized to one of 6 possible sequences of fasted or fed conditions.

Screening takes place from Day -21 to Day -1. They are admitted to the clinic on Day -1. Blood sampling for PK assessment is performed from Day 1 to Day 11 of each period. This 11 day on-site period is repeated three times in order to allow all subjects to be dosed under fed (low and high fat) and fasting conditions.

The 11 day on-site periods are separated by 7-day off site periods; subjects are checked for eligibility again one day prior to the start of a new dosing day.

Safety assessments are performed throughout the investigational period. Subjects return for an ESV at least 7 days after the last 11 day on-site period, or after withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 30.0 kg/m2, inclusive.

Exclusion Criteria:

* Known or suspected hypersensitivity to solifenacin, tamsulosin or any of the other recipients of EC905.
* Any of the contraindications or precautions for use as mentioned in the applicable sections of the Summary of Product Characteristics (SPC) of tamsulosin or solifenacin
* Use of grapefruit (more than 3 x 200 ml) or marmalade (more than three times) in the week prior to admission to the Clinical Unit, as reported by the subject.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of solifenacin by Area Under the Curve from the time of dosing until the last measurable concentration (AUClast) in plasma | Days 1-11, 18-28, 35-45
  area under the plasma concentration - time curve (AUC) from the time of dosing until the last measurable concentration (AUClast)
Pharmacokinetic parameter of solifenacin by maximum concentration (Cmax) in plasma | Days 1-11, 18-28, 35-45
  maximum concentration (Cmax)
Pharmacokinetic parameter of tamsulosin HCl by Area Under the Curve from the time of dosing until the last measurable concentration (AUClast) in plasma | Days 1-11, 18-28, 35-45
  area under the plasma concentration - time curve (AUC) from the time of dosing until the last measurable concentration (AUClast)
Pharmacokinetic parameter of tamsulosin HCl by maximum concentration (Cmax) in plasma | Days 1-11, 18-28, 35-45
  maximum concentration (Cmax)

SECONDARY OUTCOMES:
Pharmacokinetics profile of solifenacin concentration: (AUCinf), (t1/2), (tmax), (CL/F) and (Vz/F) | Days 1-11, 18-28, 35-45
  (plasma) AUC extrapolated until time = infinity (AUCinf), apparent terminal elimination half-life (t1/2), time to attain Cmax (tmax), apparent total body clearance (CL/F), apparent volume of distribution during the terminal phase (Vz/F)
Pharmacokinetics profile of tamsulosin HCl concentration: (AUCinf), (t1/2), (tmax), (CL/F) and (Vz/F) | Days 1-11, 18-28, 35-45
  (plasma) AUC extrapolated until time = infinity (AUCinf), apparent terminal elimination half-life (t1/2), time to attain Cmax (tmax), apparent total body clearance (CL/F), apparent volume of distribution during the terminal phase (Vz/F)
Safety and tolerability of single doses of EC905 (solifenacin/tamsulosin HCl) under fed or fasted conditions | Screening (Day-21 to -1) to ESV (at least 7 days after the last 11 day on-site period, or after withdrawal)
  Adverse events, clinical laboratory tests, vital signs, electrocardiogram (ECG), physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Clincial Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Parexel Early Phase Clinical Unit, Harrow, United Kingdom